CLINICAL TRIAL: NCT02160535
Title: Treatment of Chronic Post-Traumatic Headache With OnabotulinumtoxinA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to difficulty in enrolling eligible subjects
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Sylvia Lucas, Clinical Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46614
Record Dates: First submitted 2014-05-15; First posted 2014-06-10 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Chronic Post Traumatic Headache
Keywords: Mild Traumatic Brain Injury; Concussion; Post Concussive Headache
MeSH Terms: conditions — Brain Concussion | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with OnabotulinumtoxinA (Experimental): OnabotulinumtoxinA
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — 155 units of OnabotulinumtoxinA administered intramuscularly. Injections are divided across seven injection specific head/neck muscle areas every 12 weeks to prevent chronic migraine post traumatic headache
  Other Names: BOTOX

SUMMARY:
This study will provide evidence on whether the use of an FDA-approved drug therapy for the treatment of chronic migraine (OnabotulinumtoxinA) shows similar efficacy for treatment of chronic headaches caused by traumatic injury to the brain (TBI) from a direct hit to the head, or a fall, or a motor vehicle accident, or some other traumatic event.

DETAILED DESCRIPTION:
Headaches caused by trauma are called post-traumatic headaches (PTH). The Center for Disease Control estimates that between 1.4 and 1.8 million civilians in the US sustain a traumatic brain injury (TBI) each year. The objectives of the study will be evaluated in a civilian population which has sustained a mild Traumatic Brain Injury (mTBI). Research has found that the total cost due to headache in the US workforce is $20 billion per year, most of which is in the form of reduce productivity while at work. For patients with TBI who are already struggling with cognitive and health challenges in an effort to be productive, it seems reasonable to suspect that chronic PTH may slow rehabilitation efforts and successful re-entry into the work force and societal responsibility. Results from this study have the potential to contribute to recommendations for treatment of chronic PTH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild traumatic brain injury (mTBI) within the past 15 months
* Suffer at least fifteen total headache days per month
* Ability to speak and read English

Exclusion Criteria:

* Subject with hypersensitivity reactions or other intolerance to OnabotulinumtoxinA
* Previous use of OnabotulinumtoxinA for treatment of headache
* Any medications commonly used as headache preventives started less than 3 months prior to enrollment
* Prior or current diagnosis of major psychiatric disorder or other central nervous system disorder
* Less than 80% compliance (recorded for less than 24 days) in the 30 day screening headache diary
* Subjects who are pregnant or trying to become pregnant within the timeframe of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lucas, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Headache Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With OnabotulinumtoxinA
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With OnabotulinumtoxinA
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Percentage of Headache Days
Description: To measure average number of headache days three months after the last onaboltulinumtoxinA injection and compare to average number of headache days during screening month (and present as percentage of headache change).
Time Frame: Baseline, 9 months
Measure: Mean (Standard Deviation); unit: percentage of headache days
Arm/Group | Treatment With OnabotulinumtoxinA
Number analyzed (Participants) | 13
percentage of headache days
  Baseline | 83 (21)
  9 month | 49 (34)

2. Secondary Outcome: Change in SF-36 Assessment Scores
Description: Short Form-36 (SF-36) assesses quality of life. Minimum score: 0 Maximum score: 100 Higher values show improvement in quality of life.
Time Frame: Baseline and 9 month.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With OnabotulinumtoxinA
Number analyzed (Participants) | 13
score on a scale
  Baseline | 47 (30)
  9 months | 66 (29)

3. Secondary Outcome: Change in MIDAS Score
Description: Migraine Disability Assessment Minimum score: 0 Maximum score: 270 Lower values show improvement in disability.
Time Frame: Baseline and 9 month.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With OnabotulinumtoxinA
Number analyzed (Participants) | 13
score on a scale
  Baseline | 89 (51)
  9 months | 21 (18)

4. Secondary Outcome: Change in HIT-6 Score.
Description: Headache Impact Test-6 Minimum value: 36 Maximum value: 78 Lower values represent less disability.
Time Frame: Baseline and 9 month.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With OnabotulinumtoxinA
Number analyzed (Participants) | 13
score on a scale
  Baseline | 65 (4)
  9 months | 59 (7)

ADVERSE EVENTS:
Arm/Group | Treatment With OnabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With OnabotulinumtoxinA (N=13)
Increased Headache (General disorders) | 1 (1) — One subject experienced increased headache after treatment. Event thought to be local effect from injection sites and subject's sensitization to repetitive needle sticks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No